CLINICAL TRIAL: NCT06524713
Title: A 5-Year Retrospective Anesthetic Evaluation of Cases Undergoing Cesarean Section Delivery
Brief Title: A 5-Year Anesthetic Evaluation of Cases Undergoing Cesarean Section Delivery ın Our Clinic
Status: Active, not recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, sare vural yörüsün, Principal investigator, Kocaeli University
Other Study IDs: SEZRETA1822; tsahin (Other: KocaeliU)
Record Dates: First submitted 2024-01-20; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia; Cesarean Section

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite global efforts to reduce the rate of cesarean section births worldwide, increase recommendations for elective induction of labor, and promote trials of vaginal birth after previous cesarean deliveries, cesarean rates are steadily rising, varying from country to country.

The management of obstetric patients requires the effective and safe application of anesthesia to anticipate and prevent emergencies, ensuring a positive experience for the mother, baby, and their family.

Neuraxial anesthesia is considered the gold standard for cesarean section births. In case of an emergency cesarean, the likelihood of general anesthesia increases, making the safe provision of anesthesia more challenging.

The choice of anesthesia technique for cesarean section is determined by considering maternal and fetal conditions, accompanying diseases, the urgency of surgery, and the difficulty of procedures.

In this study, the investigators will retrospectively examine the anesthesia records of all cesarean section cases treated in the clinic between 2018 and 2022. the investigators aim to analyze demographic data, the anesthesia methods applied, complications, the relationship between surgery time and anesthetic method, the association between anesthesia method and neonatal Apgar scores, and the type of postoperative analgesia administered in the clinic (including regional anesthesia, opioids, non-steroidal anti-inflammatory drugs if performed). The study will be descriptive in nature, aiming to provide insights into commonly applied methods and management in the researcher's clinic.

ELIGIBILITY:
Inclusion Criteria:

* All Pregnant Women Undergoing Cesarean Section at Kocaeli University Hospital between January 1, 2018, and December 31, 2022

Exclusion Criteria:

-Ectopic Pregnancy

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant Women Undergoing Cesarean Section
Study Population: All Pregnant Women Undergoing Cesarean Section at Kocaeli University Hospital between January 1, 2018, and December 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluating the anesthetic management of cesarean section cases in researcher's clinic. | 2018-2022
  Researchers will retrospectively review patients' anesthesia records to examine anesthesia management in emergency and elective cases in the clinic.
Evaluating the anesthetic complications of cesarean section cases in researcher's clinic. | 2018-2022
  Researchers will retrospectively review patients' anesthesia records to examine common anesthesia related complications in emergency and elective cases in the clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Robson MS. Use of indications to identify appropriate caesarean section rates. Lancet Glob Health. 2018 Aug;6(8):e820-e821. doi: 10.1016/S2214-109X(18)30319-X. No abstract available. PMID 30012256
- [Background] Society of Maternal-Fetal (SMFM) Publications Committee. Electronic address: pubs@smfm.org. SMFM Statement on Elective Induction of Labor in Low-Risk Nulliparous Women at Term: the ARRIVE Trial. Am J Obstet Gynecol. 2019 Jul;221(1):B2-B4. doi: 10.1016/j.ajog.2018.08.009. Epub 2018 Aug 9. PMID 30098985
- [Background] Van de Velde M. Anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2001 Jun;14(3):307-10. doi: 10.1097/00001503-200106000-00004. PMID 17019107